CLINICAL TRIAL: NCT02155816
Title: Influence of Omega 7 + 3 Combination on Systemic Inflammation and Plasma Lipoproteins in Women: a 2-month, Double Blind, Placebo-Controlled, Randomized Community Trial
Brief Title: Omega 7 + 3 Combination and Systemic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0160
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Inflammation
Keywords: inflammation; lipoproteins; omega 3; omega 7
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): MCT (medium chain triglyceride)
  Interventions: Dietary Supplement: Placebo
- Omega 3 (Experimental): Omega-3 fatty acid ethyl esters, 2 soft gels of total 1000mg (660mg EPA +340mg DHA)/day.
  Interventions: Dietary Supplement: Omega 3
- Omega 7 + 3 (Experimental): 210mg of Omega-7 fatty acid and 1000mg (660mg EPA +340mg DHA) of Omega-3
  Interventions: Dietary Supplement: Omega 7 + 3

INTERVENTIONS:
Dietary Supplement: Omega 7 + 3 — Ingestion of omega 7 + 3 daily for 8 weeks.
  Arms: Omega 7 + 3
Dietary Supplement: Omega 3 — Omega 3 daily for 8 weeks.
  Arms: Omega 3
Dietary Supplement: Placebo — Medium chain triglycerides
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if supplementation with a mixture of omega 7 and 3 fats has a favorable influence on blood inflammation and lipoprotein biomarkers in women with systemic inflammation compared to omega 3 and placebo.

DETAILED DESCRIPTION:
Background Information and Scientific Rationale

Consumption of long-chain n-3 polyunsaturated fatty acids (n-3 PUFAs), including eicosapentaenoic acid (EPA; 20:5n-3), docosapentaenoic acid (DPA; 22:5n-3), and docosahexaenoic acid (DHA; 22:6n-3) from fish and fish-oil supplements reduces disease risk factors, counters components of the metabolic syndrome including inflammation and high triglycerides, stabilizes heart cells, prevents blood clots from forming, and decreases all-cause mortality, cardiac and sudden death, and possibly stroke (Circulation 2006;114:82-96).

The health benefits of n3-PUFAs have prompted the U.S. Food and Drug Administration (FDA) to support a qualified health claim status for EPA and DHA. Estimates are that the ratio of omega-6 (n-6) linoleic acid (LA) to omega-3 (n-3) α-linolenic acid (ALA; 18:3n-3), ALA increased from 6.4 to 10.0 during the 20th century, resulting in decreased tissue concentrations of EPA and DHA (Am J Clin Nutr 2011;93:950-962). Recommendations for EPA and DHA intake vary, but in general, most organizations recommend a range of 300 to 1,000 mg/day from fatty fish and supplements (Circulation 2006;114:82-96). The FDA recommends that consumers not exceed 3,000 mg/day of EPA and DHA, with no more than 2,000 mg/day from a dietary supplement.

The persistent increase in inflammation biomarkers is defined as chronic or systemic inflammation, and is linked with multiple disorders and diseases including atherosclerosis and cardiovascular disease (CVD), the metabolic syndrome (MetS), and diabetes mellitus (Circulation 2003;107:499-511). C-reactive protein (CRP) is the most frequently measured inflammatory biomarker, and individuals with CRP values in the upper tertile of the adult population (>3.0 mg/L) have a 2-fold increase in CVD risk compared to those with a CRP concentration below 1.0 mg/L (Curr Atheroscler Rep 2010;12:110-8). An elevated fasting IL-6 concentration is a significant component of the chronic low-grade inflammation (Metabolism 2007;56:332-8). Epidemiological studies suggest an inverse relationship between CRP and a diet rich in marine products (Am J Clin Nutr 2006;84:223-9). At sufficiently high intakes, n-3 PUFAs may decrease the production of inflammatory eicosanoids and cytokines (Mol Nutr Food Res 2008;52:885-97). The majority of intervention studies in adults with features of MetS report a benefit for some inflammatory measures, but other studies using high n-3 fatty acid doses and long supplementation periods have reported no effect (for review, see Lipids 2013;48:319-32). A pre-existing inflammatory state or a poor n-3 PUFA status may be required to see a benefit of n-3 PUFAs on systemic inflammation.

Palmitoleic acid (C16:1 n-7) is an omega-7 monounsaturated fatty acid that is found in macadamia nuts and the seeds of a variety of plants including cat's claw, sea buckthorn, and milk weed (Prog Lipid Res 2012;51:340-9). Macadamia nuts are the only practical source for palmitoleic acid (30%). The nutritional and biological functions of palmitoleic acid are complex and scientific understanding of the biological significance on human health is limited (J Lipid Res 2011;52:808-12; Curr Opin Clin Nutr Metab Care. 2013;16:225-31). Palmitoleate may increase cell membrane fluidity, attenuate insulin resistance, and reduce inflammation associated with diabetes and heart disease (for review, see Prog Lipid Res 2012;51:340-9). Several human studies indicate that supplementation and/or inclusion of macadamia nuts in a cholesterol-lowering diet significantly reduces LDL-C concentrations (4.0-10.7%) and triglyceride concentrations (9.0-20.9%) (see J Nutr 2008;138:761-7; Arch Intern Med 2000;160:1154-8). One human study with 17 male hypercholesterolemia subjects showed that supplementation with macadamia nuts for a period of 4 weeks reduced plasma biomarkers for inflammation and oxidative stress (Lipids 2007;42:583-7).

Study Product (A) Placebo Placebo (EEs)- MCT (medium chain triglyceride) and manufactured by Natural Factors. All subjects will receive one softgel orally twice daily with food.

Study Product (B): Omega-3 fatty acid ethyl esters, 2 soft gels of total 1000mg (660mg EPA +340mg DHA)/day EPA/DHA product manufactured by Natural Factors. Each softgel of Omega-3 contains 500 mg of a natural marine lipid concentrate (330 mg eicosapentaenoic acid [EPA], 170 mg docosahexaenoic acid [DHA]). All subjects will receive one softgel orally twice daily with food.

Study Product (C): Omega-3 fatty acid + Omega-7 fatty acid Cis-Palmitoleic acid, ethyl esters, 2 soft gels of total 1000mg (660mg EPA +340mg DHA) of Omega-3 + 210mg of Omega-7 fatty acid /day

All subjects will receive one soft gel orally twice daily with food.

Potential Risks and Benefits

Potential Risks of the products All of these fatty acids are found naturally in whole foods such as macadamia nuts, fish, or meat. The omega 3 supplements in this study do not exceed the upper levels recommended by the FDA (3,000 mg/day of EPA and DHA, with no more than 2,000 mg/day from a dietary supplement). For comparison, one 3-oz serving of wild Atlantic salmon provides about 1,500 mg of EPA and DHA, and a 3-oz serving of canned white tuna provides 700 mg. Fish oil supplementation has an established history of safe use as a nutritional supplement and as a medical food.

Palmitoleic acid is a monounsaturated fat that is in macadamia nuts. The purified omega 7 fat to be used in this study is derived from Peruvian anchovies, and concentrated through a seven-step purification process to 50% palmitoleic acid. In an unpublished randomized, double blinded, placebo controlled study, the omega 7 + 3 combination exerted anti-inflammatory and lipid modulating effects, and was well tolerated among participants with no adverse effects (Dr. Andrew Swick, Metagenics, private communication, February 13, 2014).

Potential Benefits Potential health benefits include improvements in plasma lipoproteins and reductions in systemic inflammation with omega 7 + 3 combination and omega 3 fats.

Study Objectives/Endpoints This is a single center, placebo controlled, double blinded, 8 week, 3-arm randomized controlled trial conducted at the Appalachian State University Human Performance Laboratory at the North Carolina Research Campus in Kannapolis, NC. All patients will undergo informed consent process before enrollment.

This is an exploratory study with generally healthy female subjects to obtain information pertaining to efficacy of omega 7 + 3 combination in improving systemic inflammation and plasma lipoproteins compared to omega 3 fats alone and placebo.

The primary Study Objectives/Endpoints are:

To explore the effects of 8-weeks supplementation with omegas 7 and 3 fats combination versus omega-3 fats and placebo on systemic inflammation (CRP and cytokine panel).

Secondary Study Objectives/Endpoints are:

To explore the effects of 8-weeks supplementation with omegas 7 and 3 fats combination versus omega-3 fats and placebo on plasma lipoproteins.

Study Design Screening/Orientation: This is a double-blinded, placebo-controlled randomized clinical study to assess the effects of placebo (A) and Omega-3 (B) and Omega-7 and Omega-3 combination (C) in the subjects. Approximately 68 female subjects between the ages of 18 and 70 years and with a BMI of 25 and higher who meet study entrance criteria will be entered into the study and randomized to one of three groups (A,B, or C). The goal is for 60 women to finish all phases of the study. The purpose of the screening/orientation visit is to determine volunteer eligibility for study participation. Screening will include review and signing of the consent form; measurement of height, weight, and body composition; completion of the medical history questionnaire and review of medical history and current medications; completion of the symptom log; and collection of 8 hour fasting blood samples for testing of CRP. Based on previous experience, approximately 100 women will have to be screened to identify 60-68 subjects with a CRP of 2 mg/L and higher. Women with a CRP below 2 mg/L will receive an email message indicating that they do not meet study criteria, but will receive results from the CRP test.

Clinical Visits:

Total length of participation in the study, including screening, will be approximately 10 weeks. Subjects will meet with the study manager at all lab visits. During the lab visits, the study manager will review questionnaires for signs and symptoms of adverse events, review compliance to the study product and lifestyle, and answer any questions from the subject. Blood samples will be collected, and body weight and composition measured at all visits. Body composition will be assessed through leg-to-leg bioelectrical impedance using a Tanita scale.

Supplement schedule: All subjects will ingest 1 soft gel (either A, B, or C) twice daily with morning and evening meals for 8 weeks. If a subject fails to ingest supplements at a given meal or day, they will be asked to double up intake to get back on schedule. Subjects failing to take supplements for three days in a row or longer will be asked to contact the research manager to review whether or not they should continue in the study. Subjects will maintain their current lifestyles - including diet, and exercise without change during trial participation. Subjects will be instructed not to make changes to their use of prescribed medications. Acetaminophen may be used as rescue for headaches and associated symptoms during study participation. The research manager will make sure the subjects are maintaining use of group A, B, or C study soft gel supplements by email between the visits. Subjects must agree to maintain normal dietary and physical activity patterns during the study, make no formal attempts to lose body weight, limit fish and seafood to no more than one serving per week, and limit intake of omega-6 fatty acids by lowering use of corn, soybean, safflower, sunflower, and similar oils, and substituting moderate amounts of olive and canola oil.

Visit 1 (Day 0) is defined as the day of enrollment and administration of the first study product. Subjects meeting all criteria including CRP levels of 2 mg/L and higher will return to the ASU-NCRC Human Performance Laboratory and receive a 28-day supply of capsules (A,B, or C). The consent form and medical questionnaire will be reviewed. A 28-day retrospective symptom log will be filled in. Weight and body composition will be assessed on the Tanita BIA scale. A blood sample will be collected, with serum sent to the Carolina Medical Center for CRP and lipid panel analysis. Plasma aliquots (EDTA tubes) will be prepared and frozen at -80°C for post-study NMR lipoprotein analysis at LipoScience (Raleigh, NC), cytokine analysis (7-plex MSD panel) at the North Carolina Research Campus, and fatty acid analysis at the Lipid Labs LLC (Austin, Minnesota).

Visit 2 (Week 4) and Visit 3 (Week 8):

Study procedures from Visit 1 will be repeated. Compliance will be assessed through the return of unused capsules.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age, female
* Body mass index (BMI) 25 kg/m2 and higher
* Generally healthy and without cardiovascular disease
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to maintain current lifestyle
* CRP values greater than or equal to 2 mg/L (established through pre-study screening).

Exclusion Criteria:

Subject Exclusion Criteria: Prohibited Medications, Medical Foods or Supplements

Exclusion criteria include the following prohibited medications, medical foods or nutritional supplements within 14 days prior to and for the duration of the study:

* Regular use of red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterol/stanol products, policosanols, or any other supplement for the control blood lipid levels.
* Use of prescription medications to control blood cholesterol and lipids including HMG Coenzyme A reductase inhibitors, bile acid sequestrants, fibrates, cholesterol adsorption blocking agents, or niacin. Common examples include Lipitor, Crestor, Zocor, Pravachol, Mevacor, Vytorin, and Niaspan.
* Regular use of omega 3 fats or fish oil medications and supplements.
* Regular use of antioxidant vitamins or supplements at doses greater than 100% Daily Value levels.
* Regular use of Aspirin and non-steroidal anti-inflammatory drugs (NSAIDs). Examples include ibuprofen (Advil, Motrin, Nuprin), naproxen (Aleve, Naprosyn), and COX-2 inhibitors (Celebrex).
* Regular use of medications classified as narcotics (e.g., codeine, Fentora, Lorcet, Vicodin, Demerol, Dolophine, OxyContin, Percocet).
* Regular use of oral or injectable corticosteroids (e.g., cortisone and prednisone).

Subject Exclusion Criteria: Medical History and Concurrent Diseases

* History of allergy or intolerance to study products including fish oils and omega-7.
* Current diagnosis or personal history of cardiovascular disease including myocardial infarction, angina, cardiovascular surgery, congestive heart failure, cardiac arrhythmias or conduction abnormalities, cerebrovascular accident, transient ischemic attack (TIA), or peripheral vascular disease, deep vein thrombosis or pulmonary embolus.
* Pregnant or planning to be pregnant during the 8-week study, or those breast feeding.

Subject Exclusion Criteria: Miscellaneous

* Inability to comply with study and/or follow-up visits.
* Any other concurrent condition which, in the opinion of the PI, would preclude participation in this study or interfere with compliance.
* Any other sound medical, psychiatric and/or social reason as determined by the PI.
* Co-enrollment in other trials is restricted other than for observational studies. Study staff should be notified of co-enrollment as it may require the approval of the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in systemic inflammation as measured with CRP and cytokines | 8 weeks
  Effects of 8-weeks supplementation with omegas 7 and 3 fats combination versus omega-3 fats and placebo on systemic inflammation (CRP and cytokine panel).

SECONDARY OUTCOMES:
Change in plasma lipoproteins (cholesterol, triglycerides, LDL-chol, HDL-chol) | 8 weeks
  Effects of 8-weeks supplementation with omegas 7 and 3 fats combination versus omega-3 fats and placebo on plasma lipoprotein panel.

CONTACTS AND LOCATIONS:
Overall Officials: David Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States